CLINICAL TRIAL: NCT04542837
Title: A Phase II Study Evaluating the Safety and Efficacy of KN046 in Combination With Lenvatinib in Advanced Hepatocellular Carcinoma
Brief Title: The Study of KN046 in Combination With Lenvatinib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Baocai Xing, Director of Surgery, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200825
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HCC
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN046 plus Lenvatinib (Experimental)
  Interventions: Biological: KN046; Drug: Lenvatinib

INTERVENTIONS:
Biological: KN046 — Subjects enrolled in the study will be intravenously administered KN046 5mg/kg every 3 weeks (Q3W), until disease progression, or unacceptable toxicity, or withdrawal of consent, or lost to follow-up, or died, or treatment for 2 years, or the investigator decides to terminate.
Drug: Lenvatinib — Subjects enrolled in the study will receive lenvatinib 12 mg (BW≥60 kg) or 8 mg (BW<60 kg) orally once a day (QD) ,until disease progression, or unacceptable toxicity, or withdrawal of consent, or lost to follow-up, or died, or treatment for 2 years, or the investigator decides to terminate.

SUMMARY:
This ia a single-arm, not-randomized, open-label phase II study. The purpose of this study is to evaluate the safety and efficacy of KN046 (PD-L1 /CTLA-4 Bispecific antibody) combined with Lenvatinib(TKI) for the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of hepatocellular carcinoma confirmed by histology or cytology；
* Barcelona Clinic Liver Cancer (BCLC) Stage B or C；
* Age ≥18 years or ≤75 years for both genders；
* ECOG performance status: 0-1；
* Child Pugh score≤7；
* LVEF≥50% or above LLN of the research institution；
* Enough organ function；
* Has at least one measurable lesion based on RECIST 1.1；
* Life expectancy ≥3 months；
* Patients must be able to understand and willing to sign a written informed consent document；

Exclusion Criteria:

* Fibrous lamina hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma etc;
* Tumor thrombus invasion at the main portal vein (Vp4), inferior vena cava or heart involvement;
* Subjects who have previously received immune checkpoint inhibitors (such as anti-PD-1/L1, CTLA-4, etc.);
* Subjects who have received liver local treatment (transcatheter chemoembolization, transcatheter embolization, hepatic artery perfusion, radiotherapy, radioembolization or ablation) within 4 weeks before administration;
* Subjects who need corticosteroids or immunosuppressive agents for systemic therapy;
* Any previous or current active autoimmune disease or history of autoimmune disease;
* History of hepatic encephalopathy or liver transplantation;
* History of interstitial lung disease or non-infectious pneumonia;
* History of allergic reactions to related drugs;
* Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients undergoing total gastrectomy;
* With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable;
* Subjects with clinically significant gastrointestinal bleeding or thrombosis or embolic events within 6 months;
* Untreated hepatitis infection: HBV DNA>2000IU/ml or10000 copies/ml, HCV RNA> 1000copy/ml, both HbsAg and anti-HCV body are positive;
* Evidence of active pulmonary tuberculosis (TB);
* Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
ORR | 1 year after the last patient's enrollment
  objective response rate (ORR) based on the RECIST 1.1 by investigator

SECONDARY OUTCOMES:
ORR | 1 year after the last patient's enrollment
  objective response rate (ORR) based on the mRECIST 1.1 and imRECIST respectively by investigator
DCR | 1 year after the last patient's enrollment
  disease control rate (DCR) based on the RECIST 1.1，mRECIST 1.1 and imRECIST respectively by investigator
DOR | 1 year after the last patient's enrollment
  duration of response (DOR) based on the RECIST 1.1，mRECIST 1.1 and imRECIST respectively by investigator
TTR | 1 year after the last patient's enrollment
  time to response (TTR) based on the RECIST 1.1，mRECIST 1.1 and imRECIST respectively by investigator
PFS | 1 year after the last patient's enrollment
OS-12m rate | 1 year after the last patient's enrollment
  12-month overall survival rate
OS | 2 year after the last patient's enrollment
  overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: Undecided